CLINICAL TRIAL: NCT00503672
Title: Assessment of Activity in Pregnancy Using an Actigraph
Status: Withdrawn | Type: Observational
Why Stopped: Data from the Actigraph devices could no longer be read/analyzed
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Deborah A. Wing, Director of Maternal Fetal Medicine, University of California, Irvine
Other Study IDs: 2006-5343
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Motor Activity; Pregnancy
Keywords: Motor Activity; Pregnancy; Accelerometer
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We would like to quantify the amount and type of activity a typical pregnant woman engages in and then compare the pregnancy outcomes of women with varying activity levels. To do this, we will have women wear a device known as an accelerometer (that records activity by measuring changes in voltage levels) at certain times in their pregnancies.

DETAILED DESCRIPTION:
General findings that have consistently been demonstrated in the literature are that activity tends to decreased during pregnancy from pre-pregnancy levels and that activity in the third trimester is less than in the first trimester. In non-pregnant patients, increase in physical activity and exercise has been associated with improved mood and self-esteem. Although the data in pregnancy is limited, available studies do suggest that inactivity is associated with worse mood. Regular physical activity is not detrimental in low-risk patients and in fact may be beneficial.

Bed rest or activity restrictions are commonly employed interventions for women with a variety of obstetric complications such as preterm contractions, vaginal bleeding, and fetal growth restriction. There is no compelling data to support bed rest as an effective therapeutic modality. There has been some data that occupational work can increase the risk of preterm birth, but other studies have not demonstrated an effect.5 Furthermore, prolonged bedrest can have detrimental effects such as muscle weakness and increased thromboembolic risk, as well as negatively impact familial relations.

The use of the accelerometer is an attempt to objectively quantify physical activity in pregnancy. The accelerometer assesses activity by measuring voltages, and can thus provide information on the intensity of activity. An additional advantage is that it can be worn on the wrist or ankle, whereas pedometers need to be worn on the waist for maximal accuracy which limits their use in pregnant women. This novel study would contribute to the existing literature on pregnancy activity that consists primarily of survey/subjective data to determine what correlation, if any, exists between activity and pregnancy outcome. Secondarily, the study will survey its participants to see if we can corroborate previous studies that have demonstrated a relationship between activity level and patients' moods.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* First trimester (11-14w)
* No medical contraindications to normal activity

Exclusion Criteria:

* Chronic medical conditions that require restricted activity (cardiac disease, severe asthma, etc)
* Known fetal anomalies
* Morbid obesity (BMI > 39)
* Maternal age less than 18 years
* Inability to comply with instructions

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant Women
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Actigraphy data points | The periods for wear have been selected such that they coincide with visits for routine prenatal screening.
  This is an observational study whose primary objective is to obtain an estimate of the amount of activity that patients engage in during a pregnancy, divided among low, moderate, and high intensity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Wing, MD, Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - Long Beach Memorial Medical Center, Miller Children's Hospital, Long Beach, California
  - University of California, Irvine, Orange, California

IPD SHARING:
Plan to Share IPD: No